CLINICAL TRIAL: NCT01078636
Title: Alzheimer's Disease Neuroimaging Initiative Grand Opportunity
Acronym: ADNI-GO
Status: Completed | Type: Observational
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: Northern California Institute of Research and Education (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IA0175; 1RC2AG036535-01 (NIH)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: amyloid; plaques; imaging; early detection; Amnestic MCI; pre-dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- EMCI (only cohort recruiting in this study): Newly recruited early amnestic Mild Cognitive Impairment patients; estimated enrollment 200
- LMCI (not recruiting in this study): Late Mild Cognitive Impairment patients; approximately 400 LMCI participants anticipated to follow from the original ADNI study
- CN (not recruiting in this study): Cognitively Normal patients; approximately 200 CN participants anticipated to follow from the original ADNI study

SUMMARY:
The purpose of this study is to build upon the information obtained in the original Alzheimer's Disease Neuroimaging Initiative (ADNI1), to examine how brain imaging technology can be used with other tests to measure the progression of mild cognitive impairment (MCI) and early Alzheimer's disease (AD). ADNI-GO seeks to define and characterize the mildest symptomatic phase of AD, referred to in this study as early amnestic MCI (EMCI). This information will aid in the early detection of AD, and in measuring the effectiveness of treatments in future clinical trials.

DETAILED DESCRIPTION:
This project continues the work from ADNI1, the goal of which is to test whether serial magnetic resonance imaging (MRI), positron emission tomography (PET), other biological markers, and clinical and neuropsychological assessments can be combined to measure the progression of mild cognitive impairment (MCI) and early Alzheimer's disease (AD). The goal of the study is to determine relationships among the clinical, cognitive, imaging, genetic, and biochemical biomarker characteristics of the stage of the AD spectrum that precedes MCI, the mildest symptomatic phase of AD, referred to here as EMCI. The ADNI-GO model posits that AD begins with amyloid β (Aβ) deposition in the cortex, which leads to synaptic dysfunction, neurodegeneration, and cognitive/ functional decline.

Some of the leading-edge technologies under study are brain-imaging techniques, such as positron emission tomography (PET), including FDG-PET (which measures glucose metabolism in the brain); PET using a radioactive compound (F-AV-45) that measures brain beta-amyloid; and structural MRI. Brain scans are showing scientists how the brain's structure and function change as AD starts and progresses. Biomarkers in cerebrospinal fluid are revealing other changes that could identify which patients with MCI will develop Alzheimer's. Scientists are looking at levels of beta-amyloid and tau in cerebrospinal fluid. (Abnormal amounts of the amyloid and tau proteins in the brain are hallmarks of Alzheimer's disease.)

All participants from ADNI1 who are in the normal and MCI stages will continue to be followed in ADNI-GO. The next step is to scan and analyze the brains of people with EMCI; 200 EMCI participants will be enrolled to narrow the gap between cognitively normal (CN) and "late MCI (LMCI)" participants currently enrolled in ADNI.

The overall impact of this study will be increased knowledge concerning the sequence and timing of events leading to MCI and AD, development of better clinical and imaging/fluid biomarker methods for early detection and for monitoring the progression of these conditions, and facilitation of clinical trials of treatments to slow disease progression, ultimately contributing to the prevention of AD.

ELIGIBILITY:
EMCI Inclusion Criteria:

* Between 55 and 90 years of age
* Study partner to accompany patient to all clinic visits for the duration of the protocol
* Memory complaint by patient and/or study partner
* Abnormal memory function score on Wechsler Memory Scale (adjusted for education)
* Mini-Mental State Exam score between 24 and 30 (inclusive)
* Clinical Dementia Rating = 0.5; Memory Box score at least 0.5
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the screening visit
* Stability of the following permitted medications for 4 weeks (unless stated otherwise):

  * Antidepressants lacking significant anticholinergic side effects
  * Estrogen replacement therapy
  * Gingko biloba is permissible, but discouraged
  * Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening
  * Cholinesterase inhibitors and memantine if stable for 12 weeks prior to screening
* Geriatric Depression Scale less than 6
* Visual and auditory acuity adequate for neuropsychological testing
* Good general health with no diseases expected to interfere with the study
* Not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile)
* Hachinski less than or equal to 4
* Six grade education or has a good work history (sufficient to exclude mental retardation)
* Fluent in English or Spanish
* Agrees to at least one lumbar puncture for the collection of CSF
* Willing and able to complete all baseline assessments
* Willing to undergo repeated MRIs and at least two PET scans and willing to provide DNA and plasma samples as specified
* Willing and able to participate in a longitudinal imaging study

Specific Inclusion Criteria for follow-up participants from ADNI1:

* Must have been enrolled and followed in ADNI for at least one year diagnosed as either Mild Cognitive Impairment (MCI) or Cognitively Normal (CN) regardless of whether a diagnostic conversion has occurred since enrolling in ADNI
* Willing and able to continue to participate in an ongoing longitudinal study; a reduced battery of tests can be requested from the project directors if the participant is not able/willing to complete the full battery
* Study partner who has frequent contact with participant and can accompany participant to all clinic visits for the duration of the protocol

Exclusion Criteria:

* Any significant neurologic disease other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
* Screening/baseline MRI scans with evidence of infection, infarction, or other focal lesions; multiple lacunes or lacunes in a critical memory structure
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body
* Major depression, bipolar disorder as described in DSM-IV within the past 1 year
* Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol
* History of schizophrenia
* History of alcohol or substance abuse or dependence within the past 2 years
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* Clinically significant abnormalities in B12, or TFTs that might interfere with the study
* Residence in skilled nursing facility
* Current use of specific psychoactive medications (e.g.,certain antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.); current use of warfarin (exclusionary for lumbar puncture)
* Use of investigational agents one month prior to entry and for the duration of the trial
* Participation in clinical studies involving neuropsychological measures being collected more than one time per year
* Exclusion for amyloid imaging with 18F -AV-45: Current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the participant in any given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1
* Exceptions to these guidelines may be considered on a case-by-case basis at the discretion of the protocol director

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Rate of Decline as measured by: Cognitive tests, Activities of Daily Living, and CDR Sum of Boxes | at screening, baseline, 6 (EMCI only) and 12 months

SECONDARY OUTCOMES:
Rate of conversion will be evaluated among all four groups | at screening , baseline, 6 (EMCI only) and 12 months
Rate of volume change of whole brain, hippocampus, and other structural MRI measures | at screening and 3, 6, and 12 months (EMCI); at baseline and 12 months (follow-up patients)
Rates of change on each specified biochemical biomarker | at baseline, 6 (EMCI only) and 12 months
Rates of change of glucose metabolism (FDG-PET) | at baseline
Extent of amyloid deposition as measured by 18F-AV-45 | at baseline
Group differences for each imaging and biomarker measurement | at screening, baseline, 6 (EMCI only) and 12 months
Correlations among biomarkers and biomarker change | at screening, baseline, 6 (EMCI only) and 12 months
Subgroups analyses: APOE genotype, low CSF Aβ42, positive amyloid imaging with 18F-AV-45 | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Petersen, MD, PhD, Study Chair — Mayo Clinic - Rochester, Minnesota; Michael W Weiner, MD, Principal Investigator — University of California, San Francisco; Paul Aisen, MD, Study Chair — University of California, San Diego
Locations (55):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, Irvine - BIC, Irvine, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Martinez, California
  - Stanford University, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wien Center, Miami Beach, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health (CCLRBC), Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Dent Neurological Group, Amherst, New York
  - New York University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital Memory & Aging Program, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas SWMC, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Canada (5):
  - University of British Columbia, Vancouver, British Columbia
  - Saint Joseph's Hospital, Hamilton, Ontario
  - Parkwood Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital / McGill University, Montreal, Quebec

REFERENCES:
- [Background] Shen L, Kim S, Risacher SL, Nho K, Swaminathan S, West JD, Foroud T, Pankratz N, Moore JH, Sloan CD, Huentelman MJ, Craig DW, Dechairo BM, Potkin SG, Jack CR Jr, Weiner MW, Saykin AJ; Alzheimer's Disease Neuroimaging Initiative. Whole genome association study of brain-wide imaging phenotypes for identifying quantitative trait loci in MCI and AD: A study of the ADNI cohort. Neuroimage. 2010 Nov 15;53(3):1051-63. doi: 10.1016/j.neuroimage.2010.01.042. Epub 2010 Jan 25. PMID 20100581
- [Background] Risacher SL, Saykin AJ, West JD, Shen L, Firpi HA, McDonald BC; Alzheimer's Disease Neuroimaging Initiative (ADNI). Baseline MRI predictors of conversion from MCI to probable AD in the ADNI cohort. Curr Alzheimer Res. 2009 Aug;6(4):347-61. doi: 10.2174/156720509788929273. PMID 19689234
- [Background] Petersen RC, Aisen PS, Beckett LA, Donohue MC, Gamst AC, Harvey DJ, Jack CR Jr, Jagust WJ, Shaw LM, Toga AW, Trojanowski JQ, Weiner MW. Alzheimer's Disease Neuroimaging Initiative (ADNI): clinical characterization. Neurology. 2010 Jan 19;74(3):201-9. doi: 10.1212/WNL.0b013e3181cb3e25. Epub 2009 Dec 30. PMID 20042704
- [Background] Misra C, Fan Y, Davatzikos C. Baseline and longitudinal patterns of brain atrophy in MCI patients, and their use in prediction of short-term conversion to AD: results from ADNI. Neuroimage. 2009 Feb 15;44(4):1415-22. doi: 10.1016/j.neuroimage.2008.10.031. Epub 2008 Nov 5. PMID 19027862
- [Derived] Miller AA, Sharp ES, Wang S, Zhao Y, Mecca AP, van Dyck CH, O'Dell RS; Alzheimer's Disease Neuroimaging Initiative (ADNI). Self-reported hearing loss is associated with faster cognitive and functional decline but not diagnostic conversion in the ADNI cohort. Alzheimers Dement. 2024 Nov;20(11):7847-7858. doi: 10.1002/alz.14252. Epub 2024 Sep 26. PMID 39324520
- See also: Laboratory of NeuroImaging: Alzheimer's Disease Neuroimaging Initiative — http://adni.loni.usc.edu/